CLINICAL TRIAL: NCT03662711
Title: Comparison of 1-year Treatment With Inhaled Long Acting Bronchodilators (LABD) Plus Inhaled Glucocorticosteroids (ICS) Versus LABD Without ICS on Re-hospitalizations and/or Death in Elderly Patients With Chronic Obstructive Pulmonary Disease (COPD) Recently Hospitalized Because of an Acute Exacerbation of COPD (ICS-Life Study).
Brief Title: Inhaled Long-acting Bronchodilators With or Without Inhaled Glucocorticosteroids for Preventing Hospitalizations and Death in Elderly Patients With Chronic Obstructive Pulmonary Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Contract terminated between AIFA and the Sponsor (University of Ferrara)
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Alberto Papi, MD, Professor, Università degli Studi di Ferrara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AIFA-ICSLIFE-001
Record Dates: First submitted 2018-08-28; First posted 2018-09-07 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: adult; drug therapy; combination; bronchodilator agents; male; female
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Bronchodilator Agents; Calcium Sulfate; GSK573719; Salmeterol Xinafoate; tiotropium-olodaterol; olodaterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long-acting beta-agonist (LABA) or LABA/LAMA (Active Comparator): long-acting bronchodilator agents (LABD, LAMA or LABA/LAMA) but no inhaled steroids plus usual care for comorbidities
  Interventions: Drug: Bronchodilator Agents
- Long-acting muscarinic antagonist (LAMA) and/or LABA plus ICS (Experimental): Bronchodilator agents LAMA and/or LABA with inhaled steroids plus usual care for comorbidities
  Interventions: Drug: Bronchodilator Agents

INTERVENTIONS:
Drug: Bronchodilator Agents — Fluticasone furoate/vilanterol
  Other Names: Revinty Ellipta
  Arms: Long-acting muscarinic antagonist (LAMA) and/or LABA plus ICS
Drug: Bronchodilator Agents — Tiotropium
  Other Names: Spiriva Respimat
  Arms: Long-acting beta-agonist (LABA) or LABA/LAMA
Drug: Bronchodilator Agents — Indacaterol
  Other Names: Onbreez Brezhaler 150
  Arms: Long-acting beta-agonist (LABA) or LABA/LAMA
Drug: Bronchodilator Agents — Umeclidinium/vilanterol
  Other Names: Laventair
  Arms: Long-acting beta-agonist (LABA) or LABA/LAMA
Drug: Bronchodilator Agents — Fluticasone propionate/salmeterol
  Other Names: Aliflus Diskus 50/500
  Arms: Long-acting muscarinic antagonist (LAMA) and/or LABA plus ICS
Drug: Bronchodilator Agents — Beclometasone dipropionate/formoterol
  Other Names: Alabaster
  Arms: Long-acting muscarinic antagonist (LAMA) and/or LABA plus ICS
Drug: Bronchodilator Agents — Budesonide formoterol
  Other Names: Fobuler
  Arms: Long-acting muscarinic antagonist (LAMA) and/or LABA plus ICS
Drug: Bronchodilator Agents — Glycopyrronium
  Other Names: Tovanor Breezhaler
  Arms: Long-acting beta-agonist (LABA) or LABA/LAMA
Drug: Bronchodilator Agents — Aclidinium
  Other Names: Bretaris Genuair
  Arms: Long-acting beta-agonist (LABA) or LABA/LAMA
Drug: Bronchodilator Agents — Umeclidinium
  Other Names: Incruse
  Arms: Long-acting beta-agonist (LABA) or LABA/LAMA
Drug: Bronchodilator Agents — Formoterol
  Other Names: Levovent
  Arms: Long-acting beta-agonist (LABA) or LABA/LAMA
Drug: Bronchodilator Agents — Indacaterol glycopyrronium
  Other Names: Ultibro Breezhaler
  Arms: Long-acting beta-agonist (LABA) or LABA/LAMA
Drug: Bronchodilator Agents — Salmeterol
  Other Names: Serevent
  Arms: Long-acting beta-agonist (LABA) or LABA/LAMA
Drug: Bronchodilator Agents — Tiotropium olodaterol
  Other Names: Spiolto Respimat
  Arms: Long-acting beta-agonist (LABA) or LABA/LAMA
Drug: Bronchodilator Agents — Aclidinium/formoterol
  Other Names: Duaklir Genuair
  Arms: Long-acting beta-agonist (LABA) or LABA/LAMA
Drug: Bronchodilator Agents — Olodaterol
  Other Names: Striverdi Respimat
  Arms: Long-acting beta-agonist (LABA) or LABA/LAMA
Drug: Bronchodilator Agents — Formoterol/glycopyrronium bromide/beclometasone dipropionate
  Other Names: Trimbow
  Arms: Long-acting muscarinic antagonist (LAMA) and/or LABA plus ICS
Drug: Bronchodilator Agents — Fluticasone furoate/umeclidinium bromide/vilanterol
  Other Names: Elebrato Ellipta
  Arms: Long-acting muscarinic antagonist (LAMA) and/or LABA plus ICS

SUMMARY:
This will be a phase IV, open label, multicenter, randomized pragmatic study in frail elderly patients with COPD. Participants will be treated with either inhaled LABD alone or LABD combined with inhaled glucocorticosteroids. The main aim of the study is to assess whether, in elderly patients with COPD and one or more cardiac comorbidities (heart failure, and/or ischemic heart disease, and/or atrial fibrillation) recently hospitalized because of an acute exacerbation of COPD, 12 months treatment with LABD(s)+ICS can increase the time to first re-hospitalization (all cause) and/or death for any cause when compared with LABD(s) alone. Patients will be followed-up for 3 months after completion of the 12 month treatment period.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease occurs mainly in the elderly and has important comorbidities, particularly cardiovascular, which increase its severity. Chronic obstructive pulmonary disease affects 5% of people globally, increasing to 10% in the elderly. According to data from the World Health Organisation (WHO), there were 384 million cases of COPD in 2010, with a global prevalence of 12% (www.who.int). Deaths due to COPD are 3 million/year globally (GOLD 2018) and >20,000/year in Italy.

The investigator speculated that multimorbid elderly COPD patients recently hospitalized due to an acute exacerbation of COPD (AECOPD) and who have concomitant cardiovascular disease may have fewer re-hospitalizations and increased survival in the following year if treated with LABD+ICS rather than with LABD alone.

The aim of this study is to examine the efficacy and safety of currently recommended and prescribed inhalation therapies to elderly, frail and multimorbid COPD patients with a recent hospitalization due to an AECOPD. The study involves a group of patients who have never before been selected for a clinical trial and who represent the 5th most common cause of hospitalization and the 3rd most common cause of death in Italy.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be older than 60 years of age, at the time of signing the informed consent.
2. Recently (within 6 months) discharged from hospital with a diagnosis of acute exacerbation of COPD (usually coded as Diagnosis Related Group (DRG) 087 or 088).
3. Participants with a clinical diagnosis of COPD (i.e. previous diagnosis of COPD and/or treatment with short acting bronchodilators (SABD), LABD or LABD+ICS
4. Spirometry confirmed diagnosis of COPD, post-bronchodilator (30 minutes after 400 μg salbutamol) FEV1/FVC ratio <0.7. The diagnostic spirometry test can have been performed up to three years prior to randomization, or if never performed before, should be performed not earlier than 4 weeks since last exacerbation
5. Smokers or ex-smokers with a smoking history of >10 pack years (a pack year is defined as 20 cigarettes smoked every day for a year)
6. Clinical diagnosis documented in the patient's medical records of one or more major chronic cardiac disease (heart failure, ischemic heart disease or atrial fibrillation).
7. Currently receiving at least one of the specified treatments (either alone or in combination, see Appendix 10.5) for heart failure, ischemic heart disease or atrial fibrillation.
8. Participant must be willing and able to perform pulmonary function tests
9. Male or female. Contraception is not considered necessary in this cohort of elderly (> 65 years) patients receiving treatment with commercially available licensed products.
10. Capable of giving signed informed consent as described in Appendix 1 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

1. Patients with a primary discharge diagnosis of DRG 087 or DRG 088 but clearly judged by the clinical investigator to be due to other causes, i.e. patients presenting to the hospital with symptoms of AECOPD but due mainly to other conditions (pulmonary embolism, pneumonia, pneumothorax, anemia, acute kidney failure, decompensated heart failure, acute ischemic heart disease, new onset atrial fibrillation, stroke, etc.)
2. Patients who required invasive mechanical ventilation during hospitalization
3. Patients with Asthma as primary and principal diagnosis
4. Patients with severe cardiovascular (CV) disease who in the opinion of the investigator are unlikely to survive the 15 month study period
5. Patients considered unable to comply with the study procedures and follow-up in the opinion of the investigator (eg, evidence of alcohol or drug abuse, psychiatric disorder, physical disability, social or geographical obstacles)
6. Patients in whom spirometry is contraindicated (eg, hemoptysis, detached retina, active tuberculosis, last trimester of pregnancy)
7. Patients with other mechanical or overt causes of respiratory symptoms, particularly dyspnea (such as pneumothorax, chest wall trauma, lung fibrosis, lung cancer, anemia, severe obesity (BMI >40) or cachexia (BMI <18))
8. Patients with any major disease which in the opinion of the investigator would prevent study participation, such as dementia, end-stage disease, cachexia, chronically bedridden patient and life expectancy <15 months.
9. Participation in any other interventional study within the last 3 months or concurrent participation in an observational clinical study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 843 (Actual)
Dates: Start 2018-11-11 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Composite event of the first time to first re-hospitalization and/or death (all cause) | 12 months

SECONDARY OUTCOMES:
Number of moderate/severe COPD exacerbations in the two patient groups | 12 months
Number of re-hospitalizations and deaths (all cause) in the two patient groups | 12 months
Quality of life (QoL) variation measured as change in COPD Assessment Test (CAT) between the two patient groups | 12 months
QoL variation measured using modified Medical Research Council (mMRC) dyspnoea scale between the two patient groups | 12 months
Number of pneumonia events | 12 months
Number of acute cardiac events | 12 months
Number of cardiovascular events | 12 months

OTHER OUTCOMES:
Change in forced expiratory volume at one second (FEV1) from baseline to the end of treatment period | 12 months
Change in forced vital capacity (FVC) from baseline to the end of treatment period | 12 months

CONTACTS AND LOCATIONS:
Locations (39):
- Italy (39):
  - Istituti Clinici Scientifici Maugeri, Pneumologia Riabilitativa, Cassano delle Murge, Apulia
  - Policlinico di Bari, U.O.C. Malattie dell'Apparato Respiratorio Universitaria, Bari, BA
  - Istituti Clinici Scientifici Maugeri S.p.A - SB, Pneumologia Riabilitativa, Telese Terme, Benevento
  - Dipartimento Di Scienze Mediche e Chirurgiche- Università Magna Grecia, Catanzaro, Calabria
  - Ospedale San Giovanni di Dio, UOC Medicina Interna, Crotone, Calabria
  - Ospedale "Jazzolino" ASP, UOC Medicina Interna, Vibo Valentia, Calabria
  - Ospedale civile di Battipaglia, Medicina, Servizio di Allergologia e Immunologia Clinica, Battipaglia, Campania
  - Azienda Ospedaliera dei Colli - Ospedale Monaldi, Napoli, Campania
  - Università degli studi di Modena e Reggio Emilia, Clinica Malattie dell'apparato Respiratorio, Modena, Emilia-Romagna
  - Azienda Ospedaliero-universitaria di Parma, Clinica pneumologica, Parma, Emilia-Romagna
  - AUSL - IRCCS di Reggio Emilia, Pneumologia, Reggio Emilia, Emilia-Romagna
  - UNIVERSITà DEGLI STUDI DI FERRARA, CLINICA DI MALATTIE DELL'APPARATO RESPIRATORIO, Ferrara, FE
  - Università degli studi di Foggia, ospedale pneumologico D'Avanzo, unità operativa di malattie dell'apparato respiratorio, Foggia, FG
  - Ospedale S. Maria degli Angeli - AAS5 Friuli Occidentale, Pneumologia, Pordenone, Friuli Venezia Giulia
  - Policlinico Universitario Campus Biomedico di Roma, Medicina Interna e Geriatria, Rome, Lazio
  - Università di Roma "Tor Vergata", Dipartimento di Medicina dei Sistemi, Malattie dell'apparato respiratorio, Rome, Lazio
  - ASL2 Savonese, Ospedale S. Corona, Pneumologia, Pietra Ligure, Liguria
  - Ospedale San Paolo, Medicina 2 e cure Intermedie, Savona, Liguria
  - Ospedale Papa Giovanni XXIII, Bergamo, Lombardy
  - Ospedale Figlie di San Camillo, Medicina Interna, Cremona, Lombardy
  - Ospedale "Carlo Poma", Struttura Complessa Pneumologia e UTIR, Mantova, Lombardy
  - Ospedale "L. Sacco" - Polo Universitario ASST Fatebenefratelli Sacco, Pneumologia, Milan, Lombardy
  - Fondazione IRCCS Policlinico San Matteo, Pneumologia, Pavia, Lombardy
  - Istituti Clinici Scientifici Fondazione Maugeri, Pneumologia Riabilitativa, Pavia, Lombardy
  - Istituti Clinici Scientifici maugeri, Pneumologia Riabilitativa, Tradate, Lombardy
  - Università degli Studi di Palermo, Ospedale "V. Cervello", Palermo, Pa
  - Ospedale Maggiore, Medicina interna, Chieri, Piedmont
  - Ospedale di Ceva, Medicina interna, San Bernardino, Piedmont
  - Ospedale Civile SS. Annunziata, Medicina interna, Savigliano, Piedmont
  - Policlinico Ospedaliero di Varese - Ospedale di Circolo e Fondazione Macchi, Medicina interna, Varese, Piedmont
  - Istituti Clinici Scientifici Maugeri, Pneumologia Riabilitativa, Veruno, Piedmont
  - Azienda Ospedaliero Universitaria "Policlinico Vittorio Emanuele", Pneumologia, Catania, Sicily
  - Ospedali Riuniti di Ancona, Pneumologia, Torrette, The Marches
  - Ospedale di Cattinara, unità operativa di pneumologia, Trieste, TS
  - Azienda Ospedaliero-universitaria Careggi, Medicina per la alta complessità Assistenziale 1, Florence, Tuscany
  - Azienda Ospedaliero-universitaria Careggi, Medicina per la alta complessità Assistenziale 2, Florence, Tuscany
  - Università degli studi di Siena, UOC Malattie respiratorie, Siena, Tuscany
  - Ospedale Cà Foncello, Treviso, Veneto
  - Ospedale Monaldi, UOC Clinica Pneumologica, Napoli

DOCUMENTS (2):
  • Study Protocol (2019-01-18): https://cdn.clinicaltrials.gov/large-docs/11/NCT03662711/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-22): https://cdn.clinicaltrials.gov/large-docs/11/NCT03662711/SAP_001.pdf